CLINICAL TRIAL: NCT00353288
Title: Comparative Study Evaluating the Immunogenicity and Safety of MeMuRu-OKA Vaccine and Measles-mumps-rubella Vaccine (Priorix™) Co-administered With Varicella Vaccine (Varilrix™) in Children Primed With Measles-mumps-rubella Vaccine
Brief Title: Immunogenicity, Safety of Measles-mumps-rubella-varicella Vaccine (MeMuRu-OKA) Compared to Priorix™ Given With Varilrix™
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 105908
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Varicella; Rubella; Measles; Mumps
MeSH Terms: conditions — Chickenpox; Rubella; Measles; Mumps

INTERVENTIONS:
Biological: MeMuRu-OKA (study vacc)
Biological: MMR, Varicella vacc (control)

SUMMARY:
As measles-mumps-rubella (MMR) vaccination is established as routine childhood practice in most industrialised countries and varicella vaccination is now being introduced in many countries during the second year of life, a combined measles-mumps-rubella-varicella vaccine was developed for administration convenience and improved compliance to vaccination. To account for situations where children have received a first dose of MMR vaccine without varicella, this study will evaluate the effect of the combined measles-mumps-rubella-varicella vaccine given in place of the second dose of MMR vaccine. A second dose of the monovalent varicella vaccine will be given to all children participating to this trial since there is a current debate on the need of a second dose to induce a full protection against varicella.

ELIGIBILITY:
Inclusion Criteria:

* Children must be healthy to participate

Exclusion Criteria:

* Immunosuppressive (including HIV) conditions, allergic diseases, neurological disorders, known anaphylactic reaction to MMR vaccine, and fever (axillary temperature ³ 37.5°C at the time of vaccination) are excluding factors.
* Children must have received one dose (but not more) of MMR at least 6 weeks before entering the study.
* They must not receive or have received other non-registered drug or vaccine within 30 days prior to study start, or immunosuppressants for more than 14 days.
* Immunoglobulins or any blood products are prohibited during the 6 months before and during the study, as well as vaccine other than that foreseen by the protocol, 30 days before until 56 days after vaccination.
* Children must not have been vaccinated against varicella.
* They must not have had measles, mumps, rubella or varicella, or have been exposed to those diseases within 30 days prior to study start.
* New-born infants (< 5 weeks of age), pregnant women without previous exposure to chickenpox, and immunodeficient persons cannot live in the same household as the vaccinated child.

Ages: 15 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 446 (Actual)
Dates: Start 2006-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Varicella seroconversion and MMR titres at 42-56 days after first vaccination

SECONDARY OUTCOMES:
Safety: solicited local/general, unsolicited AEs (42 days), SAEs (whole study)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (37):
- France (12):
  - GSK Investigational Site, Ancenis
  - GSK Investigational Site, Boulogne
  - GSK Investigational Site, Dax
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, Laon
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Lingolsheim
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Villeneuve Les Avignons
- Germany (21):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Bönnigheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Kirchzarten, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Schwieberdingen, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tettnang, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Kempten (Allgäu), Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Werneck, Bavaria
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Herford, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Neumünster, Schleswig-Holstein
- Italy (4):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Sassari, Sardinia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Gillet Y, Steri GC, Behre U, Arsene JP, Lanse X, Helm K, Esposito S, Meister N, Desole MG, Douha M, Willems P. Immunogenicity and safety of measles-mumps-rubella-varicella (MMRV) vaccine followed by one dose of varicella vaccine in children aged 15 months-2 years or 2-6 years primed with measles-mumps-rubella (MMR) vaccine. Vaccine. 2009 Jan 14;27(3):446-53. doi: 10.1016/j.vaccine.2008.10.064. Epub 2008 Nov 11. PMID 19007835
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 105908 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105908 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105908 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105908 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105908 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105908 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register